CLINICAL TRIAL: NCT01460680
Title: Association of Membrane Polyunsaturated Fatty Acid Content and Intracellular Magnesium Concentration With Mental and Physical Symptoms in Fibromyalgia and SLE: a Case-control Study
Brief Title: Membrane Polyunsaturated Fatty Acid Content in Fibromyalgia and Systemic Lupus Erythematosus (SLE)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0391-11-TLV; 0391-11 (Other: Tel Aviv Sourasky Medical Center)
Record Dates: First submitted 2011-10-10; First posted 2011-10-27 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Fibromyalgia; Systemic Lupus Erythematosus
Keywords: Fibromyalgia; Systemic Lupus Erythematosus; Omega-3 Fatty acids; Magnesium
MeSH Terms: conditions — Fibromyalgia; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Fibromyalgia patients: Patients diagnosed as suffering from Fibromyalgia according to the ACR 1990 criteria
- SLE patients: Patients diagnosed as suffering from Systemic Lupus Erythematosus by the ACR criteria
- Healthy controls: Healthy controls

SUMMARY:
Polyunsaturated omega-3 fatty acids (ω3 PUFAs) are essential nutrients. Studies indicate that the incidence of Major Depression (MD) is inversely related to the consumption of fish (which are rich in ω3-PUFAs) and to the concentration of ω3 PUFAs in the plasma or Red Blood Cell (RBC) membranes. In several studies, the ω6 to ω3 ratio was elevated (ω6 PUFAs are pro-inflammatory, compared to ω3). ω3 PUFAs are also inversely associated with anxiety and neuroticism but apparently not with somatization.

Supplementation of fish oil alleviates joint pain in patients with auto-immune disease. Inhibition of pro-inflammatory cytokines (which induce both pain and depression-like symptoms) by ω3 PUFAs may underlie the benefit conferred by fish oil consumption . RBC ω3 PUFA content is lower in patients with Systemic Lupus Erythematosus and chronic fatigue syndrome, compared to healthy controls. The ω3 PUFA status of fibromyalgia patients has not been assessed.

Magnesium is an essential nutrient and plays a regulatory role in neural transmission. It is not known whether magnesium concentration is associated with pain in humans.

The objectives of the current study are to 1) compare the mean RBC omega-3 content in female fibromyalgia patients compared to that of healthy controls and female SLE patients, and to 2) assess the correlation between RBC omega-3 content and between the severity of physical (e.g. pain) and mental (e.g. depression) in fibromyalgia and Systemic Lupus Erythematosus (SLE).

DETAILED DESCRIPTION:
Background:

Fibromyalgia is a common, chronic pai n disorder that is recognized by the American College of Rheumatology as a distinct clinical entity (1). In addition to the core feature of long-term, body-wide "soft tissue" pain, patients often report co-morbid mental and physical symptoms, including exercise intolerance, un-refreshing sleep, depressed mood and anxiety (2). Much remains to be learned from the disorder's pathophysiology, but evidence exists of inter-related perturbations involving the nervous, endocrine and immune systems (2,3). For instance, depressive and anxiety symptoms are common and frequently severe, even in community studies of FM (4). Fibromyalgia patients exhibit an increase in pro-inflammatory cytokines, which may contribute to pain and emotional distress (5,6). Although nutrients such as polyunsaturated omega-3 fatty acids and magnesium attenuate hypersensitivity to pain, little is known about the impact of nutrition on the development and persistence of fibromyalgia (7).

Polyunsaturated omega-3 fatty acids (ω3 PUFAs) are essential nutrients that are not sufficiently consumed by many individuals. The brain accrues long-chain ω3 PUFAs -particularly DHA- and a sufficient supply of ω3 PUFAs is necessary for CNS development and function (8). The accessibility of circulating PUFAs renders them suitable for assessment of PUFA status in epidemiologic studies. Indeed, studies indicate that the incidence of Major Depression (MD) is inversely related to the consumption of fish (which are rich in ω3-PUFAs) and to the concentration of ω3 PUFAs in the plasma or Red Blood Cell (RBC) membranes. RBC ω3 PUFA content is negatively correlated to the degree of depression in different settings. In several studies, the ω6 to ω3 ratio was elevated (ω6 PUFAs are pro-inflammatory, compared to ω3) (9-14). ω3 PUFAs are also inversely associated with anxiety and neuroticism (15,16) but apparently not with somatization (12).

Supplementation of fish oil alleviates joint pain in patients with auto-immune disease (17). Inhibition of pro-inflammatory cytokines (which induce both pain and depression-like symptoms) by ω3 PUFAs may underlie the benefit conferred by fish oil consumption (18). Interestingly, RBC ω3 PUFA content is lower in patients with Systemic Lupus Erythematosus (SLE, refs 19,20) and chronic fatigue syndrome (CFS, ref 21), compared to healthy controls. SLE and CFS are considered to be auto-immune and functional disorders, respectively, but both share characteristics of fibromyalgia: a higher incidence in women, increased depressive co-morbidity and the frequent presence of fibromyalgia-like symptoms (22,23). However, the ω3 PUFA status of fibromyalgia patients has not been assessed.

Magnesium is an essential nutrient and plays a regulatory role in neural transmission. It appears to counter the development of hyperalgesia by inhibition of the NMDA-receptor (24,25). Intracellular magnesium concentration reflects magnesium intake, distribution and secretion, and varies widely between individuals. It is not known whether magnesium concentration is associated with pain in humans.

The objectives of the current study are to 1) compare the mean RBC omega-3 content in female fibromyalgia patients compared to that of healthy controls and female SLE patients, and to 2) assess the correlation between RBC omega-3 content and between the severity of physical (e.g. pain) and mental (e.g. depression) in fibromyalgia and SLE.

Methods:

Study design: observational, case-control study Study Population: 100 female patients with diagnosed fibromyalgia Control population(s): 100 female SLE patients, 100 healthy adult females

Assessments: (detailed below in Procedure section):

1. Demographics and medical history
2. Body mass index
3. Mean RBC omega-3 content
4. Intracellular magnesium concentration
5. Fibromyalgia Impact Score (FIQ, bennet)
6. Modified ACR 2010 fibromyalgia scale (23)
7. Beck Depression Score
8. Pain Numeric Scale
9. SLEDAI scale (SLE patients, ref 26)

Procedure:

The study will be conducted at the Fibromyalgia Clinic (Rheumatology Unit, Sourasky Medical Center). For each patient/volunteer, all assessments (BMI, questionnaires, blood test) will be performed at a single visit. The principal investigator (K.A.) will enroll eligible and willing participants from among the female patients treated at the clinic. Eligible patients will receive a description of what is entailed in participating in the study. Suitable and willing patients will sign the informed consent form and then 1) undergo venopuncture [10 ml venous blood] and 2) complete questionnaires, with the guidance of an investigator. Data and blood samples obtained from patients will be de-identified (recoded) and stored in Clinical Research Forms (CRFs) and in test-tubes at -70oC, respectively. Blood samples will undergo fatty acid analysis (see laboratory methods) and magnesium concentration. Serum will be stored and kept for potential future analysis (e.g. for pro-inflammatory cytokines), but will not be subjected to genetic analysis.

One hundred female SLE patients treated at the Rheumatology clinic will also be enrolled. Following their signing of the informed consent form, patients will be assessed for demographic characteristics, medical history, BMI, all questionnaires, and blood analysis for RBC PUFA content and magnesium concentration. Disease activity will be documented by filling out the SLE Disease Activity Index (SLEDAI).

Healthy female volunteers (without painful or inflammatory conditions) will be enrolled through written invitation posted on allocated locations around the hospital. Following their signing of the informed consent form, volunteers will be assessed for demographic characteristics, medical history, BMI, BDI and blood analysis for RBC PUFA content and magnesium concentration.

Fatty acid composition of RBC membrane (thin liquid chromatography) 5 mls of blood will be centrifuged at 4000 rpm for 10 min at 5 o C, removal of plasma and buffy coat; addition of 5 ml cold saline + EDTA (NaCl 0.9% containing 1 mM EDTA) and mix; centrifuge at 3000 rpm for 10 min at 5oC; repeat; flushing of erythrocytes with N2; storage at -70o C (Revco). Lipid extraction will be performed by homogenization of the cells in hexane/ isopropanol (3 :2 vol./vol.) containing 5 mg/100 ml butylated hydroxytoluene as an antioxidant and 5 mg/100 ml heneicosanoic acid (21 :0) as an internal standard. Fatty acid analysis: fatty acids will be converted to methyl esters by heating with BF3 in methanol, and the methyl esters separated on a HP 5890 Series II Gas Chromatograph containing a flame ionization detector. Peak areas will be integrated and plotted with the aid of the Varian Star Integrator computer package (Varian Star Workstation, 1990, Varian Associates, Inc.). Individual fatty acid methyl esters will be identified by comparing retention times with authentic standards. Values will be expressed as wt.% of total identified fatty acids (16).

Statistical analysis:

ANOVA and Chi Square tests will be used to determine differences between the groups in possible covariates. One-way ANCOVA will be used to compare PUFA status between groups, controlling for potential covariates. Pearson correlations will be conducted (assuming a Normal distribution) to determine significant associations between symptom scores and between levels of EPA, DHA, total n-3 PUFA, AA and total n-6 PUFA (expressed in all cases as percentage of total fatty acids in erythrocytes). Significant correlations and covariates will then be entered into multiple linear regressions to investigate whether PUFA levels are associated with symptom scores. The significance level will be set at p<.05 with correction for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria (fibromyalgia):

  1. Female adults, 18-80 years old
  2. Diagnosis of fibromyalgia per ACR1990 criteria (1)

Inclusion criteria (SLE):

* Diagnosis of SLE according to the ACR criteria

Exclusion Criteria:

* Exclusion criterion (for fibromyalgia patients):

  1. Other rheumatic disease (RA, SS, symptomatic osteoarthritis etc.)
  2. Other inflammatory disease associated with musculoskeletal pain (e.g. IBD)
  3. Painful neuropathic conditions (diabetic neuropathy, post-herpetic neuralgia etc.)
  4. Pregnancy or lactation
  5. Significant fluctuation in pain level over the previous ~3 months

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 female patients attending the Fibromyalgia clinic 100 female patients diagnosed with SLE attending the rheumatology clinic 100 healthy female volunteers
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-10 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Fatty acid composition of RBC membrane | Within 2 weeks of obtaining blood sample
  5 mls of blood centrifuged at 4000 rpm for 10 min at 5 o C, removal of plasma and buffy coat; addition of 5 ml cold saline + EDTA ; centrifuge at 3000 rpm for 10 min at 5oC; repeat; flushing of erythrocytes with N2; storage at -70o C . Lipid extraction by homogenization in hexane/ isopropanol. Fatty acid analysis: fatty acids will be converted to methyl esters by heating with BF3 in methanol, and the methyl esters separated on a HP 5890 Series II Gas Chromatograph containing a flame ionization detector..

CONTACTS AND LOCATIONS:
Overall Officials: Jacob N Ablin, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center Institute of Rheumatlogy, Tel Aviv, Israel

REFERENCES:
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Arnold LM. The pathophysiology, diagnosis and treatment of fibromyalgia. Psychiatr Clin North Am. 2010 Jun;33(2):375-408. doi: 10.1016/j.psc.2010.01.001. PMID 20385343
- [Background] Maes M, Smith R, Christophe A, Cosyns P, Desnyder R, Meltzer H. Fatty acid composition in major depression: decreased omega 3 fractions in cholesteryl esters and increased C20: 4 omega 6/C20:5 omega 3 ratio in cholesteryl esters and phospholipids. J Affect Disord. 1996 Apr 26;38(1):35-46. doi: 10.1016/0165-0327(95)00092-5. PMID 8735157
- [Background] Riemer S, Maes M, Christophe A, Rief W. Lowered omega-3 PUFAs are related to major depression, but not to somatization syndrome. J Affect Disord. 2010 Jun;123(1-3):173-80. doi: 10.1016/j.jad.2009.08.004. Epub 2009 Aug 31. PMID 19720401
- [Background] Shapiro H. Could n-3 polyunsaturated fatty acids reduce pathological pain by direct actions on the nervous system? Prostaglandins Leukot Essent Fatty Acids. 2003 Mar;68(3):219-24. doi: 10.1016/s0952-3278(02)00273-9. PMID 12591006